CLINICAL TRIAL: NCT04065022
Title: The Trans-cutaneous Effects on Physiological Tremor Entertainment During tACS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Myles Mc Laughlin, Principal Investigator, KU Leuven
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: S57869-1
Record Dates: First submitted 2019-02-05; First posted 2019-08-22 (Actual); Last update posted 2019-08-22 (Actual); Status verified 2019-08

CONDITIONS: Tremor, Limb
MeSH Terms: conditions — Tremor

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Head stimulation (Experimental): Each subject will be stimulated at two different days. One day with the presence of topical anesthetic cream on the scalp above the MC and in the other day with absence of the anesthetic cream. Stimulation frequency is set similar to that of the tremor. Three stimulation amplitudes will be tested (0 mA, 0.5 mA and 2.5 mA -reduced if not uncomfortable). A set of 4*1 gel-filled cup-electrodes is placed over each of motor cortex. Each subject follows three sessions of 12 min length each day. During each session the tremor is measured while interleaving between low amplitude stimulation, high amplitude stimulation and No stimulation. By the end of each session we get 3 min of Low amplitude stimulation, 3 min of high amplitude stimulation and 6 min of No stimulation.
  Interventions: Device: tACS at tremor frequency
- Arm stimulation (Experimental): Each subject will be stimulated on only one day. Stimulation frequency is set similar to that of the tremor. Three stimulation amplitudes will be tested (0 mA, 0.5 mA and 2.5 mA -reduced if not uncomfortable). A set of 2*1 gel-filled cup-electrodes is placed over the contralateral arm. Each subject follows three sessions of 12 min length. During each session the tremor is measured while interleaving between low amplitude stimulation, high amplitude stimulation and No stimulation. By the end of each session we get 3 min of Low amplitude stimulation, 3 min of high amplitude stimulation and 6 min of No stimulation.
  Interventions: Device: tACS at tremor frequency

INTERVENTIONS:
Device: tACS at tremor frequency — tACS applied between the stimulation electrodes at tremor frequency

SUMMARY:
Transcranial alternating current stimulation (tACS) is a noninvasive neuromodulation method that works by passing alternating electric current between electrodes where at least one of them is attached to the head. This has been shown to have effects on the motor system, cognition and behavior. The exact mechanism by which tACS causes such effects is not fully understood. Some studies suggests a contribution from the stimulated peripheral nerves present in the scalp rather than direct brain effects. To test this hypothesis two arms will be done. First, 12 subjects (arm 1) will be stimulated using focused 4x1 montage with gel-filled cup-electrodes over the motor cortex and the effects will be compared between anesthetized and non-anesthetized scalp. The effects of anesthetizing the scalp will be tested on three different stimulation amplitudes off (0 mA), low (0.5 mA) and high (2.5 mA). Then, 10 subjects (arm 2) will be stimulated over the contralateral arm to exclude any direct brain stimulation effects and to test if peripheral nerve stimulation can entrain the tremor. Three outcome measurements will be measured during the experiments which are: tremor entrainment, sensation intensity and sensation threshold.

ELIGIBILITY:
Inclusion Criteria:

* Above 18
* Signed informed consents

Exclusion Criteria:

* Pregnancy
* History of Epilepsy
* Family history of Epilepsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2017-06-20 (Actual); Primary Completion 2018-01-16 (Actual); Study Completion 2018-01-16 (Actual)

PRIMARY OUTCOMES:
Change in tremor-stimulation phase entrainment- Session 1 | During session one of 12 minutes length (6 minutes with stimulation ON and 6 minutes with stimulation OFF)
  phase locking value was calculated between the tremor signal measured using accelerometer and the stimulation signal
Change in tremor-stimulation phase entrainment- Session 2 | During session two of 12 minutes length (6 minutes with stimulation ON and 6 minutes with stimulation OFF)
  phase locking value was calculated between the tremor signal measured using accelerometer and the stimulation signal
Change in tremor-stimulation phase entrainment- Session 3 | During session three of 12 minutes length (6 minutes with stimulation ON and 6 minutes with stimulation OFF)
  phase locking value was calculated between the tremor signal measured using accelerometer and the stimulation signal

SECONDARY OUTCOMES:
Sensation rating | Measured up to 5 minutes before the start of the stimulation sessions and lasts for 10 seconds of stimulation after which the subject gives the rating
  The subject is asked to rate the sensation intensity during the stimulation at each stimulation amplitude using a visual analog scale from 0 to 10. Zero means the subject doesn't feel the stimulation and the number starts to increase as the sensation perception intensity increases to reach 10 if the subject feels it painful.
Sensation threshold | Measured 3 minutes before the start of the stimulation sessions and lasts up to 2 minutes. Stimulation at each amplitude lasts for 10 seconds
  Stimulation amplitude at which the subject starts to feel the stimulation. Stimulation starts with 0 mA amplitude and then increased gradually until stimulation is perceived (or reaching maximum amplitude).

CONTACTS AND LOCATIONS:
Locations (1):
- KU Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: Undecided